CLINICAL TRIAL: NCT06762418
Title: Radiographic Analysis of Skeletal and Dentoalveolar Changes Following the Treatment of Mandibular Prognathism and Maxillary Constriction in Growing Patients Using Two Different Treatment Protocols: A Randomized Controlled Trial
Brief Title: Treating Growing Patients With Mandibular Prognathism and Maxillary Constriction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Collaborators: Universiti Sains Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-1-2025
Record Dates: First submitted 2024-12-31; First posted 2025-01-07 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Class III Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class III

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RMR with SME (Experimental): The removable mandibular retractor (RMR) will inhibit mandibular growth. This appliance will be supplemented with a medline screw that is used for slow maxillary expansion (SME).
  Interventions: Device: RMR+SME
- BAIMT with RME (Active Comparator): Bone-anchored intermaxillary traction (BAIMT) will be used for Class III correction.
  This upper part of the appliance is used for rapid maxillary expansion (RME).
  Interventions: Device: BAIMT+RME

INTERVENTIONS:
Device: RMR+SME — Patients will be asked to wear this removable appliance for 16 hours daily. The expansion screw is activated twice a week.
  Arms: RMR with SME
Device: BAIMT+RME — The elastics are worn 18 hours per day to achieve the sagittal correction. The RME appliance on the upper jaw is activated twice daily until the required expansion is achieved.
  Arms: BAIMT with RME

SUMMARY:
This randomized controlled trial intends to test the efficacy of two treatment protocols in the correction of Class III malocclusion with maxillary constriction. We have to options, either to modify the growth using inter-maxillary traction based on an upper fixed appliance that is used in the same time for rapid maxillary expansion or to inhibit mandibular growth by a removable mandibular retractor (RMR) supplied with an expansion screw.

ELIGIBILITY:
Inclusion Criteria:

1. growing male and female patients aged between 12 and 15 years
2. Angle's class III malocclusion
3. skeletal class III relationship judged clinically and confirmed radiographically (-4 < ANB < + 1)
4. An anterior crossbite involving two or more teeth or an edge-to-edge incisor relationship with or without an anterior shift of the lower jaw upon closure
5. normal inclination of the lower incisors or slightly proclined (i.e., the IMPA between 85° and 100°
6. maxillary constriction requiring expansion judged clinically and confirmed radiographically
7. permanent dentition
8. no previous orthodontic treatment

Exclusion Criteria:

1. skeletal class III malocclusion caused predominantly by maxillary deficiency (SNA<78° with a normal SNB angle)
2. severe skeletal class III presenting mainly due to mandibular protrusion (ANB < - 4° with no functional shift on closure)
3. contraindications for the use of the mini-screws, such as osteoporosis (addressed with cortisone and its derivatives) or those undergoing radiation treatment
4. a convergence between the mandibular canine root and the first premolar root ,which was assessed radiographically
5. facial asymmetry, characterized by a mandibular midline deviation exceeding 2 mm from the facial midline
6. MM angle >35° or SN-MP angle > 40°
7. The existence of cleft lip or craniofacial syndromes and/or palate abnormalities and
8. The existence of supernumerary teeth or missing ones except for the third molars.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Change in the SNA angle | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  This angle represents the position of the upper jaw in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken, and this angle will be measured in degrees.
Change in the SNB angle | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  his angle represents the position of the lower jaw in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken, and this angle will be measured in degrees.
Change in the ANB angle | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  This angle represents the relationship between the upper and lower jaws in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken, and this angle will be measured in degrees.
Change in the SN-GoMe angle | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  This angle represents the position of the lower jaw in the cephalometric analysis in the vertical direction. Lateral cephalograms will be taken, and this angle will be measured in degrees.
Change in the MM angle | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  This angle represents the amount of vertical divergence between the upper and lower jaws in the cephalometric analysis. Lateral cephalograms will be taken, and this angle will be measured in degrees.
Change in the SN-SPP angle | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  This angle represents the position of the upper jaw (represented by the spinal plane "SPP") in the vertical direction of the cephalometric analysis. Lateral cephalograms will be taken, and this angle will be measured in degrees.
Change in the Witz appraisal | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  Witz appraisal is measured by the anteroposterior distance between the projections of Points A and B onto the functional occlusal plane, measured in mm. It gives an idea about the sagittal relationship between the upper and lower jaws.
Change in the Co.Go.Me angle | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  This angle is created by the intersection between the ramus plane (Co.Go) and the mandibular plane (Go.Me). This is called the gonial angle.
Change in the mandibular length | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  This distance is measured between the mandibular condyle (Co) and the genial point (Gn).
Change in the ramus height | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  This distance is measured between the mandibular condyle (Co) and mandibular gonial angle (Go).
Change in the lower facial height | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  This distance is measured between the anterior nasal spine (ANS) and the lower point on the mandibular symphysis (Me).
Change in the A-H variable | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  This variable is the horizontal distance between A point (the maxillary bone point) and the perpendicular plane to the S-N plane through Point S (Sella).
Change in the B-H variable | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  This variable is the horizontal distance between B point (the mandibular bone point) and the perpendicular plane to the S-N plane through Point S (Sella).
Change in the SN-U1 | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  This angle represents the relationship of the upper anterior teeth with SN in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken, and this angle is going to be measured in degrees.
Change in the GoMe-L1 angle | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  This angle represents the relationship of the lower anterior teeth with the mandibular plane in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken, and this angle will be measured in degrees.
Change in the SPP-U1 angle | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  This angle represents the relationship of the upper anterior teeth with the SPP plane in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken, and this angle will be measured in degrees.
Change in ls-E Line distance | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  It is the distance between Ricketts's esthetic line and the upper lip point.
Change in li-E Line distance | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  It is the distance between the lower lip point and esthetic line of Ricketts.
Change in the Gla-Sn-Pog angle | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  It is the angle between the soft tissue forehead point (Gla) and the subnasal point (Sn) and the most anterior point on the soft tissue chin (Pog).
Change in the naso-labial angle | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  It is the angle between the upper lip and nasal columella plane.
Change in the labio-mental angle | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  It is the angle between the lower lip and the chin. It is also called the labio-mental fold angle..
Change in the Ag to MZF-j variable | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  Maxillomandibular width right: measured from the Jugal process to the frontofacial plane. This measurement is measured on the frontal cephalogram.
Change in the J-J distance | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  It is the maxillary width measured on the frontal cephalogram.
Change in the molar width at the level of apices (M-MRA) | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  This is measured between the apices of the palatal roots of the maxillary ﬁrst molars (R.RA-L.RA) on the frontal cephalogram.
Change in the molar width at the level of cusps (M-MCT) | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  This is measured between the mesio-palatal cusps tips of the maxillary ﬁrst molars (R.CT-L.CT) on the frontal cephalogram.
Change in the inferred molar tipping (M-tip) | At two assessment times: (1) one day before the beginning of the treatment, and (2) at the end of the retention phase which is expected to occur within 12 months
  The difference between R.RA-L.RA and R.CT-L.CT variables mentioned above and the difference is given in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Younis Hajeer, DDS MSc PhD, Study Director — Department of Orthodontics, Faculty of Dentistry, Damascus University, Damascus, Syria
Locations (2):
- Syria (2):
  - Adib Al-Lahham Center, Damascus Health Directorate, Ministry of Health, Damascus
  - Department of Orthodontics, Faculty of Dentistry, University of Damsacus, Damascus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Majanni AM, Hajeer MY. The Removable Mandibular Retractor vs the Bone-anchored Intermaxillary Traction in the Correction of skeletal class III Malocclusion in children: A Randomized Controlled Trial. J Contemp Dent Pract. 2016 May 1;17(5):361-71. doi: 10.5005/jp-journals-10024-1856. PMID 27443361
- [Background] Saleh M, Hajeer MY, Al-Jundi A. Assessment of pain and discomfort during early orthodontic treatment of skeletal Class III malocclusion using the Removable Mandibular Retractor Appliance. Eur J Paediatr Dent. 2013 Jun;14(2):119-24. PMID 23758461
- [Background] Saleh M, Hajeer MY, Al-Jundi A. Short-term soft- and hard-tissue changes following Class III treatment using a removable mandibular retractor: a randomized controlled trial. Orthod Craniofac Res. 2013 May;16(2):75-86. doi: 10.1111/ocr.12007. Epub 2012 Nov 8. PMID 23323964
- [Background] Rabah N, Al-Ibrahim HM, Hajeer MY, Ajaj MA. Evaluation of rapid versus slow maxillary expansion in early adolescent patients with skeletal maxillary constriction using cone-beam computed tomography: A short-term follow-up randomized controlled trial. Dent Med Probl. 2022 Oct-Dec;59(4):583-591. doi: 10.17219/dmp/133513. PMID 36108265
- [Background] Rabah N, Al-Ibrahim HM, Hajeer MY, Ajaj MA, Mahmoud G. Assessment of Patient-Centered Outcomes When Treating Maxillary Constriction Using a Slow Removable Versus a Rapid Fixed Expansion Appliance in the Adolescence Period: A Randomized Controlled Trial. Cureus. 2022 Mar 3;14(3):e22793. doi: 10.7759/cureus.22793. eCollection 2022 Mar. PMID 35261839